CLINICAL TRIAL: NCT00742287
Title: The Effects of Oligomeric Procyanidins (OPCs) on Vascular Function, Biomarkers of Oxidative Stress and Inflammation in Smokers: a Pilot Study
Brief Title: Cardiovascular Effects of Oligomeric Procyanidins (OPCs) in Smokers
Acronym: INC001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Antje Weseler, Principal Investigator, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MEC 083056
Record Dates: First submitted 2008-08-26; First posted 2008-08-27 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2011-10

CONDITIONS: Smoking
Keywords: smoking; oligomeric proanthocyanidins; polyphenols; supplementation; vascular function; oxidative stress; inflammation
MeSH Terms: conditions — Smoking; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): placebo
  Interventions: Dietary Supplement: Placebo
- 2 (Active Comparator): 200 mg oligomeric proanthocyanidins (MASQUELIER'S Original OPCs)
  Interventions: Dietary Supplement: oligomeric proanthocyanidins (MASQUELIER'S Original OPCs)

INTERVENTIONS:
Dietary Supplement: oligomeric proanthocyanidins (MASQUELIER'S Original OPCs) — 200 mg oligomeric proanthocyanidins (MASQUELIER'S Original OPCs) per day over 8 weeks
  Arms: 2
Dietary Supplement: Placebo — placebo
  Arms: 1

SUMMARY:
Smoking has been identified as a key risk factor for the development of cardiovascular diseases (CVD). It was found that a persistent increase in levels of oxidative stress and prolonged inflammation play a pivotal role in the pathogenesis of smoking associated CVD. Oligomeric proanthocyanidins (OPCs) are widely known for their anti-oxidant and anti-inflammatory effects, in vitro and in vivo. However, there are hardly any studies available that systematically investigated their acute and long-term effects on vascular function as well as on established biomarkers of oxidative stress and inflammation in an "at risk" population such as smokers.

Therefore, the aim of the present study is to investigate the effects of an eight-week supplementation with OPCs on vascular function as well as biomarkers of oxidative stress and inflammation in blood of smokers.

ELIGIBILITY:
Inclusion Criteria:

* healthy male subjects smoking ≥ 10 cigarettes per day with a regular smoking history of ≥ 5 years
* BMI ≥ 20 and ≤ 27 kg/m2

Exclusion Criteria:

* Occurence of any adverse event, in particular those which require the use of medication that might interfere with the effects and/or the uptake of the investigational products
* Intolerance of study products
* Occurence of a serious adverse event
* Use of supplements, functional foods and/or other products containing vitamins, antioxidants and polyphenolic compounds or other ingredients with potential influence on vessel function for at least one month before the beginning of the study and during the entire study
* Use of a medically prescribed diet or slimming diet
* Vegetarian or vegan lifestyle
* Excessive alcohol consumption (< 28 consumptions (approximately 250 g alcohol) per week)
* Participation in a clinical trial within 4 weeks before the study
* Non-compliance with the demands of the study

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Vasoreactivity of conduit arteries by means of flow mediated dilation (FMD) | before start of intervention and at the end of the 8 week of intervention

SECONDARY OUTCOMES:
Endothelium-dependent and -independent reactivity of microvasculature by means of Laser Doppler flowmetry (LDF) | before start of intervention, after 4 and 8 weeks of intervention
Plasma nitrite and nitrate levels | before start of intervention, after 4 and 8 weeks of intervention
Systemic oxidative stress markers such as plasma levels of PGF2alpha and TEAC, GSH erythrocyte levels and gene expression of redox enzymes | before start of intervention, after 4 and 8 weeks of intervention
Systemic inflammation markers such as plasma levels of hsCRP, fibrinogen and cytokines, as well as gene expression levels of the latter | before start of intervention, after 4 and 8 weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Antje R Weseler, PhD, Principal Investigator — Maastricht University; Aalt Bast, PhD, Prof., Study Chair — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands

REFERENCES:
- [Derived] Weseler AR, Ruijters EJ, Drittij-Reijnders MJ, Reesink KD, Haenen GR, Bast A. Pleiotropic benefit of monomeric and oligomeric flavanols on vascular health--a randomized controlled clinical pilot study. PLoS One. 2011;6(12):e28460. doi: 10.1371/journal.pone.0028460. Epub 2011 Dec 8. PMID 22174811